CLINICAL TRIAL: NCT03358667
Title: Comparison Between Dermal Matrix Membrane and Tent-screw Technique for Vertical Increase of Peri-implant Soft Tissues
Brief Title: Increase of Peri-implant Soft Tissues With Screw or Membrane
Acronym: DERMA
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the International Piezosurgery Academy, International Piezosurgery Academy
Other Study IDs: DERMA
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Alveolar Bone Loss
Keywords: peri-implant soft tissue augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — soft tissue harvesting during second stage surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: single edentulism implant insertion tent screw 2mm augmentation peri-implant soft tissue
  Interventions: Procedure: augmentation peri-implant soft tissue
- group B: single edentulism implant insertion cover screw and membrane augmentation peri-implant soft tissue
  Interventions: Procedure: augmentation peri-implant soft tissue

INTERVENTIONS:
Procedure: augmentation peri-implant soft tissue — the implant was cover with a 2 mm cover screw for a tent effect or with a dermal membrane after implant insertion

SUMMARY:
The objective of this observational study is to evaluate the growth of peri-implant soft tissues using an heterologous dermal membrane graft (group A) or a 2 mm healing screw used as a vertical support of the limbs (group B) positioned at the moment of surgical insertion of the implant.

DETAILED DESCRIPTION:
The presence of soft tissue over the implants plays an important role both in bone preservation and in enhancing aesthetic conditions. The importance of good quality and amount of soft tissues was indicated by colleagues in 1994: the soft tissue enhancement technique involved inserting, at the site of the implant, a connective tissue graft taken from the palate of the patient itself. The technique was intended to allow a better aesthetic result in the treated area and to prevent metal exposure in case of reabsorption of the vestibular bone. In a systematic review of literature, some authors in 2014 have shown that a soft tissue graft applied to the implant placement area will provide a better aesthetic result. Colleagues in 2010 tested the increase in thickness of peri-implant tissues in a randomized and controlled split-mouth study: at the time of implant placement, a site received a connective plug and one received no graft. The average thickness increase in the grafted sites was 1.3 mm and allowed for aesthetic improvement.

In recent years, some human or animal origin materials have been introduced to replace the connective tissue which, being taken by the patient, often binds to a second surgical area with increased morbidity, postoperative discomfort and longer duration of intervention same. The use of deproteinized human dermis was first introduced in plastic surgery in 1995 and ophthalmic in 1999 in the second half of the 90s and then in oral surgery. Recently colleagues used the deproteinized dermis of human origin, placed at the same time as the implants, to evaluate whether the thickening of peri-implant tissues reduced marginal bone resorption after prosthetic loading. Their study showed that areas receiving an insertion had a reduced marginal bone resorption compared to areas with thin soft tissues, without quantifying the increase in soft tissues. In another prospective study, Lorenzo and colleagues in 2011 compared the connective tissue taken from the palate to a dermal matrix of porcine origin to obtain an increase in keratinized tissue bandage: the two techniques yielded similar results. Even in this case, however, the vertical thickness increase of soft tissues was not evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. indications for implant insertion into the posterior mandible based on careful diagnosis and treatment plan;
2. presence of a residual bone crest with a minimum surgical height of 7 mm and a thickness of at least 6 mm at the programmed implant sites;
3. the bone crest must be cured (at least 6 months after the loss / extraction of the corresponding dental element);
4. Soft tissue height above the implant ≤ 2mm;
5. no regenerated bone;
6. Plaque index below 25% and bleeding index less than 20%;
7. buco-lingual amplitude of the adherent gingiva ≥ 4 mm;
8. age of the patient> 18 years;
9. patients should be able to examine and understand the study protocol;
10. informed consent.

Exclusion Criteria:

1. acute myocardial infarction in the last 2 months;
2. uncompensated coagulation turbines;
3. unmanaged diabetes (HbA1c> 7.5%);
4. head / neck district radiotherapy for the last 24 months;
5. immunocompromised patients (HIV infection or chemotherapy over the last 5 years);
6. present or past treatment with intravenous bisphosphonates;
7. psychological or psychiatric problems;
8. abuse of alcohol and / or drugs;
9. smokers

11) non-controlled periodontal disease

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: thin peri-implant biotype; one implant for one patient
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
soft tissue width | 6 months after surgery
  measurement of the full thickness flap

SECONDARY OUTCOMES:
implant survival rate | two years from surgery
  percentage of implant functional effective

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puisys A, Vindasiute E, Linkevciene L, Linkevicius T. The use of acellular dermal matrix membrane for vertical soft tissue augmentation during submerged implant placement: a case series. Clin Oral Implants Res. 2015 Apr;26(4):465-470. doi: 10.1111/clr.12401. Epub 2014 Apr 30. PMID 24779749
- [Background] Suarez-Lopez Del Amo F, Lin GH, Monje A, Galindo-Moreno P, Wang HL. Influence of Soft Tissue Thickness on Peri-Implant Marginal Bone Loss: A Systematic Review and Meta-Analysis. J Periodontol. 2016 Jun;87(6):690-9. doi: 10.1902/jop.2016.150571. Epub 2016 Jan 16. PMID 26777766